CLINICAL TRIAL: NCT02239588
Title: Evaluation of the Effect of Pure Canterbury Stage 1 Infant Formula Milk Powder on the Growth of Infant 0-6 Months of Age
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bright Dairy & Food Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 13-SC-7-BRD-002
Record Dates: First submitted 2014-09-05; First posted 2014-09-15 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-09

CONDITIONS: Growth Acceleration
MeSH Terms: interventions — Economics

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Pure Canterbury milk powder (Experimental): Oral consumption of infant formula (0-6 months) milk powder
  Interventions: Other: Oral consumption
- Other infant formula milk powder (Active Comparator): Oral consumption of milk powder (other than the experimental product) selected by subjects' parents. The products including:
  1. Yashili Ambery Infant Formula Milk Powder (Stage 1: 0-6 months)
  2. Yashili Newwit Infant Formula Milk Powder (Stage 1 0-6 months)
  3. Yashili α-golden stage Infant Formula Milk Powder (Stage 1 0-6 months)
  4. Abbott Similac Infant Formula Milk Powder (Stage 1 0-6 months)
  5. Wyeth S-26 SMA Gold Infant Formula Milk Powder (Stage 1 0-6 months)
  6. Beingmate Love plus Infant Formula Milk Powder (Stage 1 0-6 months)
  Interventions: Other: Oral consumption
- Breast milk (Placebo Comparator): Oral consumption of breast milk
  Interventions: Other: Oral consumption

INTERVENTIONS:
Other: Oral consumption — Daily oral consumption for 12 weeks:
  Placebo;
  Pure Canterbury;
  Other infant formula milk powder:
  1. Yashili Ambery Infant Formula Milk Powder (Stage 1 0-6 months)
  2. Yashili Newwit Infant Formula Milk Powder (Stage 1 0-6 months)
  3. Yashili α-golden stage Infant Formula Milk Powder (Stage 1 0-6 months)
  4. Abbott Similac Infant Formula Milk Powder (Stage 1 0-6 months)
  5. Wyeth S-26 SMA Gold Infant Formula Milk Powder (Stage 1 0-6 months)
  6. Beingmate Love plus Infant Formula Milk Powder (Stage 1 0-6 months)

SUMMARY:
This was a randomized, double-blind, single-center, placebo-controlled, three-arm study, with a 12-week intervention period.

The objectives of this study were to evaluate the effect of Pure Canterbury Stage 1 (0-6 months) milk powder on:

1. Bone health;
2. Infants growth;
3. Intestinal health;
4. Gastrointestinal tolerance to the test product;

g) Incidence of Eczema

DETAILED DESCRIPTION:
• Quality control of the study: 1.1 Study monitoring and source data verification: Monitoring was done according to the monitoring plan by a representative of the investigator, who checked the case report forms for completeness and clarity, and cross-checked them with source documents. In addition to the monitoring visits, frequent communications (letter, telephone, fax, e-mail), by the study monitor ensured that the investigation was conducted according to protocol design and regulatory requirements. Study close-out was performed by the study monitor upon closure of the study.

1.2 On-site audits: Domestic and foreign regulatory authorities, the IEC/IRB, and an auditor authorized by the sponsor may request access to all source documents, case report forms, and other study documentation for on-site audit or inspection. Direct access to these documents was guaranteed by the investigator, who must provide support at all times for these activities. Medical records and other study documents may be copied during audit or inspection provided that subject names are obliterated on the copies to ensure confidentiality.

1.3 Documentation: A case report form was provided for each subject. All protocol-required information collected during the study was entered by the investigator, or designated representative, in the case report form. Details of case report form completion and correction were explained to the investigator.

The investigator, or designated representative, should complete the case report form pages as soon as possible after information is collected, preferably on the same day that a study patient is seen for an examination, treatment, or any other study procedure. Any outstanding entries must be completed immediately after the final examination. An explanation should be given for all missing data.

A source data location list was prepared prior to study initiation. This list was filed in both the trial master file and the investigator study file and updated as necessary.

The completed case report forms were reviewed and signed by the investigator named in the clinical study protocol or by a designated sub investigator.

The sponsor would retain the original of all completed case report forms. The principal investigator kept the copies of all completed case report forms for 25 years after the trial based on Good Clinical Practice (GCP) requirements.

• Quality assurance of study products: All products used in this study were manufactured and provided by Bright Dairy & Food Co., Ltd. The quality test of study products was conducted by Shanghai dairy products quality supervision and inspection station. The study products were stored at the study site and assigned to the subjects by the investigator. The amount of products received and assigned were filed on product distribution list by the investigator. The study products were not allowed to be given to anyone who didn't participated in the study. No sales of unassigned products was allowed. After the completion of the study, the unassigned products need to be returned to Bright Dairy & Food Co., Ltd.

The products were labeled with study code. A master participation list was completed which identifies each patient full name and unique identification number. The identity of the specific product was blind to patients, support staff and investigators. The unmasking occurred to the investigators and statistical analyses team only after completion of statistical analyses.

• Data management: Study data were recorded on Case Report Forms (CRFs) and then entered into saved in the form of Excel files. Data was double entered and cross-validated.

• Management of subject withdrawal: A number of 120 subjects were enrolled in the study.

Subjects may be withdrawn from the study for the following reasons:

* At their own request or at the request of their legally authorized representative,
* If, in the investigator's opinion, continuation in the study would be detrimental to the patient's well-being,
* If they are lost to follow-up. In all cases, the reason for and date of withdrawal must be recorded in the Exit Form and in the subject's medical records and the sponsor's representative must be notified within 5 days. The subject must be followed up to establish whether the reason was an adverse event, and, if so, this must be reported in accordance with the procedure of an adverse event (described bellow). The investigator must make every effort to contact subject lost to follow-up. Attempts to contact such subject must be documented in the subject's records (e.g., dates and times of attempted telephone contact).

Investigator must be notified of all serious or unexpected adverse events within 48 hours. Notification does not depend on whether there is a connection to the study formula or not. All adverse events must be documented on the appropriate pages of the case report forms.

• Statistical analysis plan: Analysis was performed for the intent-to-treat population. Chi-square test was used comparison among study groups for categorical data. For continuous outcomes, one-way ANOVA was used for between-group comparison, followed by multiple comparison with Bonferroni adjustment. Paired t-test was used for pre-post comparison within each study group. Non-parametric methods were used for non-normal data, data with unequal variances. The analysis was completed using the statistical package SPSS17.0.

ELIGIBILITY:
Inclusion Criteria:

* Infants 7~90 days old;
* Fed by breast milk before enrollment;
* Concent form signed by parents

Exclusion Criteria:

* Twins, multiple births, low birth weight children, over birth weight children or early birth children with gestational age less than 37 weeks;
* During pregnancy, the mothers had pregnancy complications or other disease that may affect the study results;
* Having serious diseases that may affect study interventions, such as neonatal sepsis, pneumonia (associated with respiratory failure), heart failure and other diseases;
* Having neonatal diarrhea or acute respiratory infections within 48 hours before enrollment;
* Having potential metabolic diseases, chronic diseases, congenital malformations, central nervous system disorders, neuromuscular disorders or diseases affecting bone metabolism that may affect growth or the study results;
* Having taken any food containing prebiotics or probiotics within 15 days of enrollment;
* Having gluten allergy (celiac disease);
* Body weight-to-height Z-value <-3 according to the standard of WHO;
* Receiving hormone therapy and intravenous nutrition;
* Lactose intolerance;
* Have participated in other clinical studies within 3 months prior to the date of screening;
* Unable to comply the study schedule

Ages: 7 Days to 90 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2014-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Bone density change from baseline (Tibial speed of sound measurement) | After 12 weeks of study intervention
  Week 12 values minus Baseline (week 0) values

SECONDARY OUTCOMES:
Growth measurements | Baseline (week 0), week 4, week 8, week 12
  Body weight (g), Height (cm), Head circumference (cm), Chest circumference (cm),
Stool consistency | Daily up to 12 weeks
Fecal short-chain fatty acid concentration | Baseline (week 0), week 12
Fecal bacteria count | Baseline (week 0), week 12
  Bifidobacteria Lactobacteria Clostridium perfringens
Intestinal adherence questionnaire | Daily up to 12 weeks
Incidence of Eczema | Baseline (week 0), week 4, week 8, week 12
Adverse event | Daily up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyang Sheng, MD, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- XinHua Hospital Affiliated to Shanghai JiaoTong University, Shanghai, China